CLINICAL TRIAL: NCT04465279
Title: Evaluation of Trifocal Diffractive Intraocular Lens After Cataract Extraction With Phacoemulsification
Brief Title: Trifocal Diffractive Intraocular Lens After Cataract Extraction With Phacoemulsification
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0000755
Record Dates: First submitted 2020-06-28; First posted 2020-07-10 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-06

CONDITIONS: Refractive Errors
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Intervention Model Description: This is a prospective, non-comparative, non-randomized study including 36 eyes had implantation of trifocal diffractive IOL
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trifocal Diffractive Intraocular Lens (FineVision) (Experimental): 36 eyes having implantation of trifocal diffractive IOL (FineVision)
  Interventions: Device: Trifocal diffractive intraocular lens

INTERVENTIONS:
Device: Trifocal diffractive intraocular lens — Trifocal IOL having foldable single-piece fully diffractive pupil dependent aspheric IOL. Which have been made of hydrophilic acrylic with an ultraviolet (UV) and blue light inhibitor. It has an optic diameter of 6.15 mm and an overall diameter of 10.75 mm; it has +3.5D additional power for near vision and +1.75 D additional power for intermediate vision, consisting of 26 diffractive steps.
  Other Names: (FineVision IOL)

SUMMARY:
Multifocal IOLs that maintain distance focus and improve near vision have been developed to reduce spectacle dependence.Multifocal IOLs improve patient performance of near-vision tasks, such as reading crafts, hobbies, and social activities to a greater extent than do monofocal IOLs. However, halos and reduced contrast sensitivity have been associated with multifocal IOLs and are common reasons for patient's dissatisfaction.Trifocal technology has been developed to create intermediate focus to overcome these difficulties. Continuous reports of the visual outcomes of the FineVision trifocal IOLs are encouraging.

DETAILED DESCRIPTION:
Monofocal IOLs, which provide effective distance vision, currently account for the majority of IOLs implantations. Patients who have undergone cataract surgery with implantation of monofocal IOL may require spectacles to perform near-distance (e.g., reading) or intermediate-distance (e.g., using a computer) tasks depending on their visual demandsMultifocal IOLs that maintain distance focus and improve near vision have been developed to reduce spectacle dependence.Multifocal IOLs improve patient performance of near-vision tasks, such as reading crafts, hobbies, and social activities to a greater extent than do monofocal IOLs. However, halos and reduced contrast sensitivity have been associated with multifocal IOLs and are common reasons for patient's dissatisfaction.Trifocal technology has been developed to create intermediate focus to overcome these difficulties. Continuous reports of the visual outcomes of the FineVision trifocal IOLs are encouraging.

ELIGIBILITY:
Inclusion Criteria:

* patient eyes had cataract with no other pathology, patients desire for spectacle independence after surgery and with realistic expectation.

Exclusion Criteria:

* Any ocular comorbidity that affect the end results of the surgery, history of ocular trauma, irregular corneal astigmatism, pupil abnormalities and capsular or zonular abnormalities that may affect postoperative centration as tilt of the lens (e.g. pseudo exfoliation syndrome and Marfan's syndrome).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Visual Acuity | 3 months
  Current study used Sloan chart (Good - Lite Co, USA) for intermediate, Snellen chart for far and Landolt ring chart for near vision
Defocus curve | 3 months
  examined monocular and binocular after correcting distant VA refractive error then inserting defocus lenses 0.50-D focus steps from (+1.50 to -3.50 D) in the trial frame

SECONDARY OUTCOMES:
Contrast sensitivity | 3 months
  using the CSV-1000 contrast test.
Visual Satisfaction Questionnaire | 3 months
  Questionnaire patient satisfaction protocol mediated by (PhysIOL Lige, Belgium).

CONTACTS AND LOCATIONS:
Overall Officials: Ehab Mossallam, PhD, Principal Investigator — Alexandria Faculty of Medicine
Locations (1):
- Alexandria Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zein El-Dein AA, Elmassry A, El-Hennawi HM, Mossallam EF. Objective and subjective evaluation of trifocal diffractive intraocular Lens after cataract extraction with phacoemulsification: a prospective clinical study. BMC Ophthalmol. 2021 Apr 14;21(1):179. doi: 10.1186/s12886-021-01937-z. PMID 33849466